CLINICAL TRIAL: NCT06859684
Title: Hepatic Arterial Infusion Chemotherapy (HAIC) Combined With Durvalumab and Lenvatinib in Patients With Locally Advanced or Metastatic Intrahepatic Cholangiocarcinoma: a Phase 2 Study(HAIC-quad Trial)
Acronym: HAIC-quad
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Wen Tianfu, Director of Liver Surgery Department, West China Hospital, Sichuan University, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAIC-quad-01
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-02

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc); HAIC; Durvalumab
Keywords: locally advanced or metastatic intrahepatic cholangiocarcinoma; durvalumab; Lenvatinib; HAIC
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension | interventions — durvalumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HAIC-quad Arm (Experimental)
  Interventions: Drug: Durvalumab; Drug: hepatic arterial infusion chemotherapy (HAIC); Drug: Lenvatinib

INTERVENTIONS:
Drug: Durvalumab — Durvalumab: During combination therapy: 1500 mg, Q3W, during combination therapy, on days 3-5 of each 3-week cycle (determined by the investigator); during maintenance therapy: 1500 mg Q4W
Drug: hepatic arterial infusion chemotherapy (HAIC) — hepatic arterial infusion chemotherapy (HAIC) : GemCis regimen was adopted, with the specific regimen as follows: cisplatin 60 mg/m2 on the first day, arterial infusion for half an hour, gemcitabine 1000 mg/m2 on the first day, arterial infusion for half an hour, repeated once every 3 weeks, and 4-6 cycles of treatment (the specific number of cycles was determined by the investigator according to the patient's condition).
Drug: Lenvatinib — Lenvatinib 8mg (weight <60 kg) or 12mg (weight ≥60 kg) oral QD, during combination therapy, starting on day 3 of each 3-week cycle (determined by the investigator)

SUMMARY:
At present, the first-line treatment for patients with advanced unresectable intrahepatic cholangiocarcinoma is mainly systemic treatment, but the improvement in efficacy is limited and is not enough to meet the current clinical treatment needs. Hepatic artery infusion chemotherapy (HAIC) has the advantages of increasing local drug concentration and reducing toxic side effects compared to systemic intravenous chemotherapy. In order to enable patients with advanced intrahepatic cholangiocarcinoma to obtain better treatment effects, this study plans to explore HAIC combined with durvalumab and lenvatinib as the first-line treatment for patients with locally advanced or metastatic ICC, in order to provide a better treatment choice for their comprehensive treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed intrahepatic cholangiocarcinoma, with a preliminary diagnosis of unresectable or metastatic disease and no previous systemic treatment.

   Anatomical factors: ① Patients with invasion of the portal vein, hepatic vein or main bile duct, who cannot undergo resection and reconstruction; ② Patients with decompensated cirrhosis or severe portal hypertension, and the residual liver FLR does not meet the safe liver resection decision-making system Biological factors: ① Multiple tumors in the left and right livers; ② Metastasis to distant lymph nodes such as the para-aorta or distant organ metastasis
2. Disease recurrence > 6 months after radical surgery; if adjuvant therapy is given after surgery, patients > 6 months after completion of adjuvant therapy (chemotherapy and/or radiotherapy) are eligible for inclusion.
3. WHO/ECOG PS of 0 or 1
4. There was at least 1 target lesion (TL) that met the RECIST 1.1 criteria

Exclusion Criteria:

1. Patients who have received systemic treatment in the past.
2. Patients with severe liver dysfunction (Child-Pugh C grade), or significant jaundice, hepatic encephalopathy, refractory ascites, or hepatorenal syndrome.
3. Patients with severe and uncorrectable coagulation dysfunction.
4. Patients with active hepatitis or severe infection who cannot be treated simultaneously.
5. Patients with cachexia or multiple organ failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 26 months
  Disease assessments based on investigator assessments were determined by using RECIST version 1.1 guidelines. The ORR was defined as the percentage of patients with confirmed complete response (CR) or confirmed partial response (PR). The CR was defined as disappearance of all target and non-target lesions and no new lesions. The PR was defined as >= 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new non-target lesion. A confirmed CR or PR was defined as 2 CRs or 2 PRs with no evidence of progression in-between. Patients who discontinued randomized treatment without progression, received a subsequent anti-cancer therapy and then responded were not included as responders for ORR.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 36 months
  Overall Survival (OS) was defined as the time from the date of randomization until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique.
Progression-free Survival (PFS) | Up to approximately 26 months
  PFS based on investigator assessments according to RECIST version 1.1 was defined as time from date of randomization until date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdrew from randomized therapy or received another anticancer therapy prior to progression. Progression (i.e., PD) was defined as at least a 20% increase in the sum of diameters of target lesions (TLs) and an absolute increase of ≥5mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters, or a measurable increase in a non-target lesion, or the appearance of new lesions. Median PFS was calculated using the Kaplan-Meier technique.
Number of Participants Who Experience One or More Adverse Events (AE) | Up to approximately 36 months
  An adverse event (AE) was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided